CLINICAL TRIAL: NCT02528747
Title: A Multi-Center Observational Survey of Breast Cancer Patients With Metastatic Bone Disease Receiving Oral Ibandronate (BONDORAL)
Brief Title: A Survey of Breast Cancer Patients With Metastatic Bone Disease Receiving Oral Ibandronate
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22421
Record Dates: First submitted 2015-08-06; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Study population: Breast cancer patients with metastatic bone disease

SUMMARY:
This observational, multicenter survey is designed to assess the efficacy of oral ibandronate in adults with breast cancer and metastatic bone disease. Data on the use of ibandronate in clinical practice will be collected from Hungarian patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Histologically confirmed breast cancer with bone metastasis
* Receiving or indicated for the tablet formulation of ibandronate according to the summary of product characteristics (SmPC) and local labeling

Exclusion Criteria:

* Contraindication to ibandronate according to SmPC
* Ongoing participation in any trial evaluating the efficacy and/or safety of ibandronate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with metastatic bone disease who are receiving oral ibandronate will be followed for approximately 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in bone pain according to Visual Analog Scale (VAS) score | From Baseline to the end of 1 year

SECONDARY OUTCOMES:
Compliance with tablet formulation of ibandronate according to Case Report Form (CRF) questionnaire | Up to approximately 1 year
Incidence of adverse events | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Hungary (18):
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Kaposvár
  - Kecskemét
  - Kistarcsa
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Veszprém
  - Zalaegerszeg